CLINICAL TRIAL: NCT03112681
Title: A Phase 2, Prospective, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate Safety, Tolerability and Efficacy of Saroglitazar Magnesium in Patients With Primary Biliary Cholangitis (EPICS )
Brief Title: Study to Evaluate Safety, Tolerability and Efficacy of Saroglitazar Mg in Patients With Primary Biliary Cholangitis
Acronym: EPICS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zydus Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SARO.16.004
Record Dates: First submitted 2017-04-10; First posted 2017-04-13 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Primary Biliary Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — saroglitazar

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Saroglitazar magnesium 2 mg (Experimental): Saroglitazar magnesium 2 mg tablet Once daily for 16 weeks
  Interventions: Drug: Saroglitazar magnesium 2 mg
- Saroglitazar magnesium 4 mg (Experimental): Saroglitazar magnesium 4 mg tablet Once daily for 16 weeks
  Interventions: Drug: Saroglitazar magnesium 4 mg
- Placebo (Placebo Comparator): Placebo tablet Once daily for 16 weeks
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Saroglitazar magnesium 2 mg — Saroglitazar magnesium 2 mg once daily in the morning before breakfast without food, for a period of 16 weeks.
  Other Names: Not any
  Arms: Saroglitazar magnesium 2 mg
Drug: Saroglitazar magnesium 4 mg — Saroglitazar magnesium 4 mg once daily in the morning before breakfast without food, for a period of 16 weeks.
  Other Names: Not any
  Arms: Saroglitazar magnesium 4 mg
Drug: Placebo Oral Tablet — Placebo once daily in the morning before breakfast without food, for a period of 16 weeks.
  Other Names: Not any
  Arms: Placebo

SUMMARY:
prospective, multicenter, randomized, double-blind, placebo-controlled study to evaluate safety, tolerability and efficacy of saroglitazar magnesium 2 mg, 4 mg in Patients with Primary Biliary Cholangitis (PBC). A total 36 subjects will be enrolled in a ratio of 1:1:1 to receive either saroglitazar magnesium 2 mg or saroglitazar magnesium 4 mg or placebo.

DETAILED DESCRIPTION:
Study SARO.16.004.02 is a prospective, multicenter, randomized, double-blind, placebo-controlled study to evaluate safety, tolerability and efficacy of saroglitazar magnesium 2 mg, 4 mg in Patients with Primary Biliary Cholangitis.

A total 36 subjects will be enrolled in a ratio of 1:1:1 to receive either saroglitazar magnesium 2 mg or saroglitazar magnesium 4 mg or placebo. The primary objective is to investigate the effect of a 16-week treatment regimen of Saroglitazar magnesium 2 mg and 4 mg on alkaline phosphatase (ALP) levels in patients with Primary Biliary Cholangitis.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, between 18 and 75 years of age, inclusive.
2. a) Patients on therapeutic doses of Ursodeoxycholic acid (UDCA) for ≥12 months and stable therapy for ≥3 months prior to enrolment.

   OR b) Patients who are unable to tolerate UDCA, and did not receive UDCA for at least 3 months from the date of screening.
3. History of confirmed Primary Biliary Cholangitis Diagnosis, based on American Association for the Study of Liver Disease [AASLD] and European Association for Study of the Liver [EASL] Practice Guidelines; [Lindor 2009; EASL 2009], as demonstrated by the presence of at least≥2 of the following 3 diagnostic factors:

   * History of elevated Alkaline Phosphatase levels for at least 6 months prior to Screening Visit 1
   * Positive antimitochondrial antibodies (AMA) titer or if AMA negative or in low titer (<1:80) PBC specific antibodies (anti-GP210 and/or anti-SP100 and/or antibodies against the major M2 components [PDC-E2, 2-oxo-glutaric acid dehydrogenase complex])
   * Liver biopsy consistent with PBC.
4. ALP ≥1.67x upper limit of normal (ULN) at Visit 1 and Visit 2 and with < 30% variance between the levels from Visit 1 to Visit 2.
5. Contraception: Female patients must be postmenopausal, surgically sterile, or if premenopausal, agree to use ≥ 1 effective method of contraception during the trial. Effective methods of contraception are considered to be Hormonal (e.g., contraceptive pill, patch, intramuscular implant or injection); or Double barrier method, i.e., (a) condom (male or female) or (b) diaphragm, with spermicide; or Intrauterine device (IUD); or Vasectomy (partner).
6. Must provide written informed consent and agree to comply with the trial protocol.

Exclusion Criteria:

1. Consumption of >3 units of alcohol per day (>21 units per week) if male and >2 units of alcohol per day (>14 units per week) if female for at least 3 consecutive months in the last 5 years (Note: 1 unit = 12 ounces of beer, 4 ounces of wine or 1 ounce of spirits/hard liquor).
2. History or presence of other concomitant liver diseases including:

   * Hepatitis B or C virus (HCV, HBV) infection
   * Primary sclerosing cholangitis (PSC)
   * Alcoholic liver disease
   * Definite autoimmune liver disease or overlap syndrome
   * Non-alcoholic steatohepatitis (NASH)
3. Cirrhosis with complications, including history or presence of: spontaneous bacterial peritonitis, hepatocellular carcinoma, bilirubin > 2x ULN, ascites, encephalopathy, known esophageal varices or history of variceal bleeding and active or history of hepatorenal syndrome.
4. History of any venous thromboembolism, transient ischemic attack (TIA), intracranial hemorrhage, neoplasm, arteriovenous malformation, vasculitis, bleeding disorder, coagulation disorders or screening blood tests that indicate altered coagulability (e.g. platelet count, activated partial thromboplastin time [aPTT], partial thromboplastin time [PTT] or thrombin time [TT] tests).
5. Patients with INR > upper limit of normal (ULN) at visit 1.
6. Patients with total bilirubin > ULN at visit 1 that is not due to Gilbert's syndrome
7. Patients with >30% increase in ALT, total bilirubin, or Internation normalized ratio (INR) between Visit 1 to Visit 2.
8. Patients with serum creatinine >ULN according to the gender at Visit 1.
9. Patients with abnormal total creatine kinase (CK) OR lipase OR amylase at Visit 1.
10. Unstable cardiovascular disease, including:

    * unstable angina, (i.e., new or worsening symptoms of coronary heart disease within the past 3 months), acute coronary syndrome within the past 6 months, acute myocardial infarction in the past 3 months or heart failure of New York Heart Association class (III - IV) or worsening congestive heart failure, or coronary artery intervention, within the past 6 months
    * history of (within prior 3 months) or current unstable cardiac dysrhythmias
    * uncontrolled hypertension (systolic blood pressure [BP] >160 mmHg and/or diastolic BP >100 mmHg)
    * stroke or transient ischemic attack within the prior 6 months
11. History of malignancy in the past 5 years and/or active neoplasm with the exception of resolved superficial nonmelanoma skin cancer.
12. Contraindications to Saroglitazar magnesium or has any conditions affecting the ability to evaluate the effects of Saroglitazar magnesium.
13. Known allergy, sensitivity or intolerance to the study drug, comparator or formulation ingredients.
14. Participation in any other clinical study within the previous 3 months of screening.
15. Illicit substance abuse within the past 6 months.
16. History or other evidence of severe illness or any other conditions that would make the patient, in the opinion of the investigator, unsuitable for the study (such as poorly controlled psychiatric disease, human immunodeficiency virus (HIV), coronary artery disease or active gastrointestinal conditions that might interfere with drug absorption).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-08-18 (Actual); Primary Completion 2020-08-07 (Actual); Study Completion 2020-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deven Parmar, MD FACP FCP, Study Director — Zydus Therapeutics Inc.
Locations (9):
- United States (9):
  - California Liver Research Institute, Pasadena, California
  - Schiff Center for Liver Diseases/University of Miami, Miami, Florida
  - Gastrointestional Specialists of Georgia, Marietta, Georgia
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Rutgers NJ Medical School, Newark, New Jersey
  - Carolinas Healthcare System, Charlotte, North Carolina
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Einstein Medical Center Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Background] European Association for the Study of the Liver. EASL Clinical Practice Guidelines: management of cholestatic liver diseases. J Hepatol. 2009 Aug;51(2):237-67. doi: 10.1016/j.jhep.2009.04.009. Epub 2009 Jun 6. No abstract available. PMID 19501929
- [Background] Lindor KD, Gershwin ME, Poupon R, Kaplan M, Bergasa NV, Heathcote EJ; American Association for Study of Liver Diseases. Primary biliary cirrhosis. Hepatology. 2009 Jul;50(1):291-308. doi: 10.1002/hep.22906. No abstract available. PMID 19554543
- [Result] Vuppalanchi R, Caldwell SH, Pyrsopoulos N, deLemos AS, Rossi S, Levy C, Goldberg DS, Mena EA, Sheikh A, Ravinuthala R, Shaikh F, Bainbridge JD, Parmar DV, Chalasani NP. Proof-of-concept study to evaluate the safety and efficacy of saroglitazar in patients with primary biliary cholangitis. J Hepatol. 2022 Jan;76(1):75-85. doi: 10.1016/j.jhep.2021.08.025. Epub 2021 Sep 4. PMID 34487750
- [Derived] Vuppalanchi R, Gonzalez-Huezo MS, Payan-Olivas R, Munoz-Espinosa LE, Shaikh F, Pio Cruz-Lopez JL, Parmar D. A Multicenter, Open-Label, Single-Arm Study to Evaluate the Efficacy and Safety of Saroglitazar in Patients With Primary Biliary Cholangitis. Clin Transl Gastroenterol. 2021 Mar 26;12(4):e00327. doi: 10.14309/ctg.0000000000000327. PMID 33769355
- See also: European Association for the Study of the Liver. EASL Clinical Practice Guidelines: management of cholestatic liver diseases. — http://pubmed.ncbi.nlm.nih.gov/19501929/
- See also: Lindor KD, Gershwin ME, Poupon R, Kaplan M, Bergasa NV, Heathcote EJ; American Association for Study of Liver Diseases. Primary biliary cirrhosis. — http://pubmed.ncbi.nlm.nih.gov/19554543/
- See also: Vuppalanchi R, Caldwell SH, Pyrsopoulos N, deLemos AS, Rossi S, Levy C, Goldberg DS. Proof-of-concept study to evaluate the safety and efficacy of saroglitazar in patients — http://pubmed.ncbi.nlm.nih.gov/34487750/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg | Placebo
Started | 14 | 13 | 10
Completed | 13 | 10 | 9
Not Completed | 1 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg | Placebo | Total
Number analyzed (Participants) | 14 | 13 | 10 | 37
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.21 (9.67) | 55.08 (8.00) | 59.20 (7.30) | 57.00 (8.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 10 | 36
  Male | 1 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 0 | 4
  Not Hispanic or Latino | 10 | 12 | 10 | 32
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 3
  White | 13 | 11 | 9 | 33
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.71 (6.39) | 29.62 (6.49) | 32.30 (7.37) | 29.62 (6.77)

OUTCOME MEASURES:

1. Primary Outcome: Effect of a 16-week Treatment Regimen of Saroglitazar Magnesium 2 mg and 4 mg on Alkaline Phosphatase (ALP) Levels in Patients With Primary Biliary Cholangitis.
Description: Change in ALP levels after 16 weeks of Saroglitazar magnesium 2 mg and 4 mg treatment.
Time Frame: Baseline and Week 16
Population: Modified intent-to-treat population
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 14 | 13 | 10
U/L | -163.82 (111.84) | -162.31 (113.98) | -11.15 (27.36)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 2 mg vs Placebo; Test type: Superiority; p = 0.0001, paired t-test
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Test type: Superiority; p = 0.0002, paired t-test

ADVERSE EVENTS:
Time Frame: 16 Weeks
Arm/Group | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13 | 0/10
Serious Adverse Events (participants affected / at risk) | 2/14 | 0/13 | 0/10
Other Adverse Events (participants affected / at risk) | 12/14 | 11/13 | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Saroglitazar Magnesium 2 mg (N=14) | Saroglitazar Magnesium 4 mg (N=13) | Placebo (N=10)
Oedema peripheral (General disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Saroglitazar Magnesium 2 mg (N=14) | Saroglitazar Magnesium 4 mg (N=13) | Placebo (N=10)
Nausea (Gastrointestinal disorders) | 1 | 2 | 1
Constipation (Gastrointestinal disorders) | 2 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 0
Herpes Zoster (Infections and infestations) | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 1
Inflammation (General disorders) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2
Hepatic Enzyme increased (Investigations) | 0 | 2 | 0
Transaminase increased (Investigations) | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypervitaminosis D (Metabolism and nutrition disorders) | 0 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 1
Abdominal distention (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 1 | 0
Anal Pruritus (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal Motility Disorder (Gastrointestinal disorders) | 0 | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Oedema peripheral (General disorders) | 1 | 1 | 0
Oedema (General disorders) | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Biopsy skin (Investigations) | 0 | 1 | 0
Liver function test increased (Investigations) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0
Vestibular migraine (Nervous system disorders) | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Blepharal pigmentation (Eye disorders) | 0 | 1 | 0
Eye irritation (Eye disorders) | 0 | 1 | 0
Retinal tear (Eye disorders) | 0 | 0 | 1
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0
Stress urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-08-21): https://cdn.clinicaltrials.gov/large-docs/81/NCT03112681/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-11): https://cdn.clinicaltrials.gov/large-docs/81/NCT03112681/SAP_001.pdf